CLINICAL TRIAL: NCT01611363
Title: An Exploratory Study to Investigate the Effects of Ipragliflozin (ASP1941) on Glucose Homeostasis and Urinary Glucose Excretion in Healthy Subjects and Subjects With Type 2 Diabetes Mellitus (T2DM)
Brief Title: A Phase 1 Study to Investigate the Mechanism of Action of Ipragliflozin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1941-CL-0050; 2010-024070-19 (EudraCT Number)
Record Dates: First submitted 2012-05-31; First posted 2012-06-05 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Ipragliflozin; Phase 1; Healthy; Diabetes Mellitus; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — ipragliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A (Experimental): Ipragliflozin (low dose) & Placebo
  Interventions: Drug: ASP1941; Drug: Placebo
- Part B (Experimental): Ipragliflozin (high dose)
  Interventions: Drug: ASP1941

INTERVENTIONS:
Drug: ASP1941 — Oral
  Other Names: Ipragliflozin
Drug: Placebo — Oral
  Arms: Part A

SUMMARY:
In this study the effect of ipragliflozin on glucose homeostasis in healthy subjects and T2DM subjects, and the effect of exposure of ipragliflozin on urinary glucose excretion and plasma glucose in T2DM subjects will be investigated.

DETAILED DESCRIPTION:
This study will consist of 2 parts. In Part A the effect of ipragliflozin on the glucose homeostasis will be investigated and in Part B we will investigate the effect of exposure of ipragliflozin on UGE and plasma glucose levels.

Part A

This part will be a randomized, double-blind, placebo-controlled, 2-

period, 2 treatment crossover design in healthy subjects and in T2DM

subjects who are drug naïve or washed out for metformin prior to

admission to the clinical site.

Part B

This part will be an open-label, randomized, 2-period, 2 treatment

crossover design in T2DM subjects stratified by baseline HbA1c

levels (6.0-6.9%, 7.0-7.9%, 8.0-8.9% or 9.0-9.9%).

ELIGIBILITY:
Inclusion Criteria:

Inclusion Part A: Healthy subjects

* Subject is healthy without diabetes mellitus
* Subject has a fasted plasma glucose (FPG) of less than 5.6 mmol/l at screening
* Subject has a Body Mass Index (BMI) more than or equal to 18.5 and less than 28.0 kg/m2
* Subject's serum creatinine is within the normal range

Inclusion Part A: T2DM subjects

* Subject has been diagnosed with T2DM for at least 6 months
* Subject's body mass index (BMI) is equal to or more than 20.0 and less than 35.0 kg/m2 at screening
* Subject has a HbA1c level above 7.0% and less than 9.0% at screening
* Subject has a (FPG) of less than 10.0 mmol/l
* Subject is treatment naïve to glucose-lowering medication or uses metformin that will be washed out at least 3 weeks prior to the first dosing at Day 1
* Subject's serum creatinine is within the normal range

Inclusion Part B: T2DM subjects

* Subject has a body mass index (BMI) of more than or equal to 20.0 and less than 35.0 kg/m2 at screening.
* Subject has been diagnosed with T2DM for at least 6 months
* Subject has HbA1c level of equal to or more than 6.0% and less than 10% at screening
* Subject has a FPG of less than 10.0 mmol/l
* Subject is drug naïve or on a stable glucose lowering therapy (metformin, TZD, DPP-4 inhibitor or SUD therapy

Exclusion Criteria:

Exclusion Part A: Healthy subjects

* Any of the liver function tests above the upper limit of normal
* A QTc interval of >430 ms (males) and >450 ms (females), a history of unexplained syncope, cardiac arrest, unexplained significant cardiac arrhythmias or torsades de pointes, structural heart disease, or a family history of Long QT Syndrome (LQTS)
* Abnormal pulse and/or blood pressure measurements at screening as follows: Pulse <40 or >90 bpm; mean systolic blood pressure >140 mmHg; mean diastolic blood pressure >90 mmHg
* eGFR (based on Modification of Diet in Renal Disease (MDRD) method) less than 60 ml/min/1.73m2 on Day -2

Exclusion Part A & Part B: T2DM subjects

* Subject has type 1 diabetes mellitus
* A QTc interval of >450 ms (males) and >470 ms (females), a history of unexplained syncope, cardiac arrest, unexplained significant cardiac arrhythmias or torsades de pointes, structural heart disease, or a family history of Long QT Syndrome (LQTS)
* Subject is on an insulin therapy or has received insulin within 3 months prior to screening, with the exception of acute use of <7 days prior to screening
* Subject has a urinary microalbumin/creatinine ratio above or equal to 300 mg/g at screening
* Subject has an ALT and/or AST higher than 3 times the upper limit of normal or has a total bilirubin more than 2 times the upper limit of normal at screening
* Subject has a symptomatic urinary tract infection or symptomatic genito-urinary infection at screening
* Subject has persistent, uncontrolled severe hypertension as indicated by a mean systolic blood pressure > 160 mmHg or a mean diastolic blood pressure of > 100 mmHg
* Subject has significant cardiovascular disease
* eGFR (based on MDRD method) less than 60 ml/min/1.73m2 on Day -2

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-10-27 (Actual); Primary Completion 2012-02-03 (Actual); Study Completion 2012-02-03 (Actual)

PRIMARY OUTCOMES:
Part A: Assessment of glucose homeostasis in fasted condition and after an oral glucose load, following multiple doses of ipragliflozin in healthy subjects and subjects with T2DM | 4 days
Part A: Assessment of peripheral glucose utilization after an oral glucose load, following multiple doses of ipragliflozin | 4 days
Part A: Assessment of splanchnic uptake after an oral glucose load, following multiple doses of ipragliflozin | 4 days
Part A: Assessment of mean glucose levels in fasted condition and after an oral glucose load, following multiple doses of ipragliflozin | 4 days
Part B: Assessment of the relationship between the exposure to ipragliflozin in plasma, urinary glucose excretion and plasma glucose levels in subjects with T2DM | 6 days (PK), 12 days (urine) and 8 days (PD)

SECONDARY OUTCOMES:
Part A: Assessment of steady state urinary sodium excretion and urinary glucose excretion following multiple doses of ipragliflozin | 4 days (sodium) and 14 days (glucose) days
Part A: Assessment of energy production and utilization of energy sources following multiple doses of ipragliflozin | 4 days
Part A: Safety and tolerability following multiple doses of ipragliflozin assessed by recording adverse events, laboratory assessments, vital signs, electrocardiograms (ECGs) and signs and symptoms of hypoglycemia | Up to 21 days
Part B: Safety and tolerability following multiple doses of ipragliflozin assessed by recording adverse events, laboratory assessments, vital signs, electrocardiograms (ECGs) and signs and symptoms of hypoglycemia | Up to 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Director — Astellas Pharma Europe B.V.
Locations (1):
- Neuss, Germany

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=4